CLINICAL TRIAL: NCT05819671
Title: Prevalence of Upper Limb Musculoskeletal Abnormalities in Type 2 Diabetic Patients and Its Relation to Glycemic Control.
Brief Title: Prevalence of Upper Limb Musculoskeletal Abnormalities in Type 2 Diabetic Patients and Its Relation to Hypoglycemic Control.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eslam Elsayed Ali Shohda (Other Government)
Responsible Party: Sponsor-Investigator, Eslam Elsayed Ali Shohda, General Committee of Teaching Hospitals and Institutes, Egypt, General Committee of Teaching Hospitals and Institutes, Egypt
Organization: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Other Study IDs: HAH00016
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2022-12

CONDITIONS: Upper Limb Musculoskeletal Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Groupe(A): Group (A)diabetics - g
- group(B): group B normal is a normal control(non-diabetics)

SUMMARY:
to investigate prevalence of upper limb musculoskeletal disorders and correlations to glycemic control.

DETAILED DESCRIPTION:
). DM is associated with a number of complications including renal disease, peripheral neuropathy, retinopathy, vascular events and musculoskeletal complications. DM is complicated by musculoskeletal problems of upper extremity and particularly the hand, collectively referred as "the diabetic hand." (3) The most common upper limb musculoskeletal disorders associated with DM are adhesive capsulitis, rotator's cuff tendinitis, limited joint mobility (LJM), Dupuytren's disease (DD), trigger finger (TF), and carpal tunnel syndrome (CTS). Upper limb musculoskeletal disorders affect hand functions and activities of daily living (ADL). Aim of the study: to investigate prevalence of upper limb musculoskeletal disorders and correlations to glycemic control.

Inclusion criteria: patients will be included to this study(cases) if they are:

1) Diabetic patients. 2) Age > 18 years. 3) Diagnosed as type 2.

Exclusion criteria:

Patients will be excluded if they have rheumatoid arthritis, other rheumatological diseases or previous upper limb surgeries.

Sample size calculation: By reviewing literature, it is found that the most relevant study (3) to our work found that the prevalence of upper limb musculoskeletal abnormalities in type 2 diabetic patients is .22 and for control group is .05 so, by using piface calculator (version 1.76) to calculate sample size (power = 0.8, alpha error = 0.05 and beta= 0.2) it is found that we need 71 participants for every group. To increase power of the study will enroll 100 participants for every group.

ELIGIBILITY:
Inclusion Criteria:

* patients will be included to this study(cases) if they are: 1) Diabetic patients. 2) Age > 18 years. 3) Diagnosed as type 2.

Exclusion Criteria:

- Patients will be excluded if they have rheumatoid arthritis, other rheumatological diseases or previous upper limb surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetics type 2 - comparable control
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of upper limb musculoskeletal disorders and correlations to glycemic control | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Dr Shohda, hd,pt, Principal Investigator — GOTHI
Locations (1):
- Al ahrar teaching hospital, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No
data only for study researchers and the organization under which the study is conducted